CLINICAL TRIAL: NCT01084135
Title: A 20-Week Double-Blind Placebo Controlled Clinical Trial to Evaluate the Safety and Efficacy of Rivastigmine in Children (Ages 10-18) With Down Syndrome
Brief Title: Rivastigmine Study in Adolescents With Down Syndrome
Acronym: DS-Riv
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Taishoff Family Foundation (Unknown); Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00013682
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2015-03-12 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-02

CONDITIONS: Down Syndrome
Keywords: Clinical trial; Down syndrome; adolescents; cognitive; rivastigmine
MeSH Terms: conditions — Down Syndrome | interventions — Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rivastigmine- Liquid form (Experimental): At the baseline visit (week 0), the subject will begin rivastigmine treatment at a dose of 0.75 mg bid. This dose will be continued for two weeks and then increased to 1.5 mg bid for an additional eight weeks. At the week 10 safety visit, the dose will be increased to 4.5 mg/day (3.0 mg and 1.5 mg) for an additional 10 weeks. If a subject is unable to tolerate a particular dose, the dose will be lowered to the previously tolerated dose, down to a minimum of 0.75 mg bid. If the subject is unable to tolerate the 0.75 mg bid dose he/she will be dismissed from the study.
  Interventions: Drug: Rivastigmine
- Liquid placebo (Placebo Comparator): Subjects receiving placebo will maintain matched titration volume increase as treatment arm. The placebo will be matched to liquid rivastigmine in consistency and taste.
  Interventions: Other: Liquid Placebo

INTERVENTIONS:
Drug: Rivastigmine — At the baseline visit (week 0), the subject will begin rivastigmine treatment at a dose of 0.75 mg bid. This dose will be continued for two weeks and then increased to 1.5 mg bid for an additional eight weeks. At the week 10 safety visit, the dose will be increased to 4.5 mg/day (3.0 mg and 1.5 mg) for an additional 10 weeks. Subjects receiving placebo will maintain the same schedule. If a subject is unable to tolerate a particular dose, the dose will be lowered to the previously tolerated dose, down to a minimum of 0.75 mg bid. If the subject is unable to tolerate the 0.75 mg bid dose he/she will be dismissed from the study.
  Other Names: Rivastigmine-Excelon
  Arms: Rivastigmine- Liquid form
Other: Liquid Placebo — Subjects receiving placebo will maintain matched titration volume increase as treatment arm. The placebo will be matched to liquid rivastigmine in consistency and taste.
  Arms: Liquid placebo

SUMMARY:
The purpose of this study is to determine if short term use of rivastigmine can improve functional abilities (for example, language, memory, and executive function) in adolescents with Down syndrome.

DETAILED DESCRIPTION:
This 24 week, double-blind, placebo controlled trial will be completed at the Clinical Research Unit of Duke University Medical Center and at the Kennedy Krieger Institute (KKI). Sixteen evaluable subjects will be enrolled at Duke and 24 evaluable subjects will be enrolled at KKI. The study consists of four visits, a screening visit (-4 weeks), a baseline visit (week 0); a safety visit at week 10, and a final/termination visit at week 20.

The specific aims of this study are to: a) investigate efficacy of rivastigmine tartrate treatment; b) build upon our open-label treatment results of overall function and language improvement in adolescents with Down syndrome (DS) in a double-blind, placebo-controlled clinical trial; and c) investigate other specific cognitive domains that may selectively respond to rivastigmine tartrate treatment.

The original IRB-approved protocol included the Parent/Caregiver Rating Form of the Vineland Adaptive Behavior Scales- Second Edition (VABS-II) . The protocol was amended to replace the Parent/Caregiver Rating Form of the Vineland Adaptive Behavior Scales- Second Edition (VABS-II) with the Vineland Adaptive Behavior Scales, Second Edition, Survey Interview Form. The protocol was also amended to extend the trial from 12 weeks to 20 weeks. Due to the changes in the amended protocol the subject enrolled prior to the IRB amendment will not be included in the data analysis section.

ELIGIBILITY:
Inclusion Criteria:

1. Correct VERBAL responses for 7/9 of the Expressive One Word Picture Vocabulary Test items.
2. Subject able to put at least 2-3 words together in conversational speech.
3. Subject's speech is understandable to the examiner for the majority of the time.
4. Subjects are in good health and medically stable

Exclusion Criteria:

1. Subject uses sign language as a primary means of communication
2. Subject has a medical history that contraindicate the use of rivastigmine (For example, patients with active seizure disorders, asthma, celiac disease, heart disease or heart rhythm disorders).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2009-11; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kishnani, MD, Principal Investigator — Duke University; George Capone, MD, Principal Investigator — Kennedy Krieger Institute/Johns Hopkins
Locations (2):
- United States (2):
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Duke University Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 participant started and completed the 12 week period. The protocol was amended and 23 subject enrolled into the 20 week amended period (22 completed).
Pre-assignment Details: 42 subjects signed consent, 10 were screen failures, 1 withdrew consent prior to being assigned to an arm, 1 was withdrawn by PI after being assigned an arm for noncompliance, 30 completed study.
Period: 12 Week
Arm/Group | Rivastigmine- Liquid Form | Liquid Placebo
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0
Period: 20 Week
Arm/Group | Rivastigmine- Liquid Form | Liquid Placebo
Started | 12 | 11
Completed | 12 | 10
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- 20 Week Rivastigmine- Liquid Form: At the baseline visit (week 0), the subject will begin rivastigmine treatment at a dose of 0.75 mg bid. This dose will be continued for two weeks and then increased to 1.5 mg bid for an additional eight weeks. At the week 10 safety visit, the dose will be increased to 4.5 mg/day (3.0 mg and 1.5 mg) for an additional 10 weeks. If a subject is unable to tolerate a particular dose, the dose will be lowered to the previously tolerated dose, down to a minimum of 0.75 mg bid. If the subject is unable to tolerate the 0.75 mg bid dose he/she will be dismissed from the study.
- 20 Week Liquid Placebo; 12 Week Liquid Placebo: Subjects receiving placebo will maintain matched titration volume increase as treatment arm. The placebo will be matched to liquid rivastigmine in consistency and taste.
  Liquid Placebo: Subjects receiving placebo will maintain matched titration volume increase as treatment arm. The placebo will be matched to liquid rivastigmine in consistency and taste.
- 12 Week Rivastigmine- Liquid Form: At the baseline visit (week 0), the subject will begin rivastigmine treatment at a dose of 0.75 mg bid. This dose will be continued for two weeks and then increased to 1.5 mg bid for an additional four weeks. At the week 6 safety visit, the dose will be increased to 4.5 mg/day (3.0 mg and 1.5 mg) for an additional 6 weeks.
- Total: Total of all reporting groups
Arm/Group | 20 Week Rivastigmine- Liquid Form | 20 Week Liquid Placebo | 12 Week Rivastigmine- Liquid Form | 12 Week Liquid Placebo | Total
Number analyzed (Participants) | 12 | 11 | 4 | 4 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 11 | 4 | 4 | 31
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 2 | 2 | 18
  Male | 4 | 5 | 2 | 2 | 13
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 4 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Vineland Adaptive Behavior Scales, Second Edition (Survey Interview Form)
Description: The Vineland Adaptive Behavior Scales, Second Edition (Survey Interview Form) is a measure of adaptive behavior in children, adolescents and adults. It yields an overall standard score (Adaptive Behavior Composite, ABC) and age standard scores in four domains. ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160). Higher scores suggest a higher level of adaptive functioning. In this study, the change between each subject's ABC at Baseline and the Final Visit was computed. A rise in standard scores from Baseline to the Final Visit indicates improvement.
Time Frame: Baseline & Study termination (Week 20)
Population: All subjects who completed the 20 week period were included in analysis except for 2 subjects whose form was completed incorrectly.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine- Liquid Form | Liquid Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | -1.7 (3.2) | 2.0 (3.6)

2. Secondary Outcome: Behavior Rating Inventory of Executive Function-Preschool (BRIEF-P)
Description: The Behavior Rating Inventory of Executive Function-Preschool Version (BRIEF-P) is a parent report measure of executive function behaviors in children in their home setting. It yields an overall score (Global Executive Composite, GEC) that is based on its five clinical scales. Raw scores range from 63 to 189. Higher scores suggest that an individual's executive function skills are more problematic. In this study, the change between each subject's raw score at Baseline and the Final Visit was computed for the Global Executive Composite. A decline in raw scores from Baseline to the Final Visit indicates improvement.
Time Frame: Baseline and Final (Week 20) visit
Population: All subjects who completed the 20 week period were included in analysis except for 1 subjects whose form was completed incorrectly.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rivastigmine- Liquid Form | Liquid Placebo
Number analyzed (Participants) | 11 | 10
units on a scale | -3.6 (7.7) | -6.1 (12.0)

ADVERSE EVENTS:
Groups:
- 20 Week: Rivastigmine- Liquid Form: At the baseline visit (week 0), the subject will begin rivastigmine treatment at a dose of 0.75 mg bid. This dose will be continued for two weeks and then increased to 1.5 mg bid for an additional eight weeks. At the week 10 safety visit, the dose will be increased to 4.5 mg/day (3.0 mg and 1.5 mg) for an additional 10 weeks. If a subject is unable to tolerate a particular dose, the dose will be lowered to the previously tolerated dose, down to a minimum of 0.75 mg bid. If the subject is unable to tolerate the 0.75 mg bid dose he/she will be dismissed from the study.
- 20 Week: Liquid Placebo; 12 Week: Liquid Placebo: Liquid Placebo: Subjects receiving placebo will maintain matched titration volume increase as treatment arm. The placebo will be matched to liquid rivastigmine in consistency and taste.
- 12 Week: Rivastigmine- Liquid Form: At the baseline visit (week 0), the subject will begin rivastigmine treatment at a dose of 0.75 mg bid. This dose will be continued for two weeks and then increased to 1.5 mg bid for an additional four weeks. At the week 6 safety visit, the dose will be increased to 4.5 mg/day (3.0 mg and 1.5 mg) for an additional 6 weeks.
Arm/Group | 20 Week: Rivastigmine- Liquid Form | 20 Week: Liquid Placebo | 12 Week: Rivastigmine- Liquid Form | 12 Week: Liquid Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 11/12 | 8/11 | 3/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 Week: Rivastigmine- Liquid Form (N=12) | 20 Week: Liquid Placebo (N=11) | 12 Week: Rivastigmine- Liquid Form (N=4) | 12 Week: Liquid Placebo (N=4)
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 0 | 3
Nausea (Gastrointestinal disorders) | 3 | 3 | 1 | 1
Stomach ache (Gastrointestinal disorders) | 5 | 3 | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 1 | 0
Trouble sleeping (Nervous system disorders) | 1 | 1 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Shakiness (Nervous system disorders) | 0 | 1 | 0 | 0
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumps in neck (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Boil (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Menstural cramps (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Cut (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Restless legs (Nervous system disorders) | 1 | 0 | 0 | 0
Pale coloring (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Foot twitching (Nervous system disorders) | 1 | 0 | 0 | 0
Itchy (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Eye twitch (Eye disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Increased bilirubin (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Indigestion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Worsening acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Cold (General disorders) | 3 | 2 | 0 | 0
Stomach flu (General disorders) | 2 | 0 | 0 | 0
Fever (General disorders) | 0 | 2 | 0 | 0
Worsening alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Leg cramps (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 1 | 1 | 0 | 0
Assertive, stubborn, more emotional (Psychiatric disorders) | 1 | 0 | 0 | 0
Fainted (Nervous system disorders) | 1 | 0 | 0 | 0
Sleepy (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Frequent urination (Renal and urinary disorders) | 0 | 1 | 1 | 0
Weight gain (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
excessive gas (Gastrointestinal disorders) | 0 | 0 | 1 | 0
behavior problems (Psychiatric disorders) | 0 | 0 | 3 | 1
Vaginal yeast infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary track infection (Renal and urinary disorders) | 0 | 1 | 0 | 0
nightmares (Psychiatric disorders) | 0 | 0 | 1 | 0
acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No